CLINICAL TRIAL: NCT06515691
Title: Evaluation of Effectiveness of Ultrasound-Guided Modified Thoracoabdominal Nerve Plane Block Through Perichondrial Approach (M-TAPA) for Postoperative Analgesia Management in Patients Undergoing Laparoscopic Sleeve Gastrectomy Operation
Brief Title: Modified Thoracoabdominal Nerve Plane Block In Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ayse Ince, Assist Prof, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 3
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Bariatric Surgery; Laparoscopic Sleeve Gastrectomy; Acute Post Operative Pain
Keywords: ModifiedThoracoabdominal Nerve Plane Block; Laparoscopic Sleeve Gastrectomy; Bariatric Surgery; Acute Postoperative Pain
MeSH Terms: conditions — Obesity; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Sixty patients aged 18-65 years old with American Society of Anesthesiologists (ASA) classification II-III, scheduled for laparoscopic sleeve gastrectomy operation will be included in the study. Patients will be randomly divided into two groups (Group M=M-TAPA block group, Group K = control group) including 30 patients each, before entering the operating room.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcomes assessor and participants will be blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M = M-TAPA Block group (Experimental): M-TAPA block will be performed andd standard postoperaive pain management protocols will be applied.
  Interventions: Procedure: M-TAPA block; Procedure: Postoperative pain management
- Group K = control group (Active Comparator): Standard postoperative pain management protocols will be applied. No plane block will be applied.
  Interventions: Procedure: Postoperative pain management

INTERVENTIONS:
Procedure: M-TAPA block — After the wound closure is completed and the patient is still under genaral anesthesia the M-TAPA block ill be performed. As the patient is in the supine position, the high-frequency linear US probe (11-12 MHz, Vivid Q) and a 22-G 80-mm needle (Stimuplex® Ultra 360®, Braun, USA) will be placed in a sagittal position at the costochondral junction at the level of the 9th and 10th ribs. After the rib and the external oblique, internal oblique, and transversus abdominis muscles are visualized on USG, using an in-plane technique, the block needle will be advanced and the block location will be confirmed by injecting 5 ml of saline between the internal oblique and transversus abdominis muscles. Once the block location is confirmed, 30 ml of 0.25% bupivacaine (Buvicaine ®) will be applied on each side. The total volume will be 60 ml.
  Arms: Group M = M-TAPA Block group
Procedure: Postoperative pain management — ibuprofen 400mg (Ibuprofen-PF®) intravenous (IV), and tramadol (Contramal®) 100 mg IV will be administered to all patients 20 minutes before wound closure. After surgery, Ibuprofen 400 mg will be given three times a day. A patient-controlled analgesia (PCA) system containing 10 mcg/ml fentanyl will be provided to all patients without continuous infusion. Patients can administer boluses of 0.35 mcg/kg with a 15-minute lockout period and a maximum dose of 100 mcg per hour. Another anesthesiologist will assess patients after surgery. If the patient's pain score (NRS) is 4 or higher, IV tramadol (Contramal®) 100 mg will be given as a rescue analgesic.

SUMMARY:
Ultrasound-guided Modified Thoracoabdominal Nerve Plane Block (M-TAPA) is performed into the costochondral aspect at the 9th-10th costal level by injecting local anesthetics deep into the chondrium. It provides blockage of both the anterior and lateral cutaneous branches of the thoracoabdominal nerve. Studies show that M-TAPA block is effective for postoperative analgesia and other abdominal surgeries, but its effect on patients undergoing LSG surgery has not yet been studied. The hypothesis is that the M-TAPA block performed in patients undergoing Laparoscopic Sleeve Gastrectomy (LSG) Operation would reduce opioid consumption in the first 24 hours period after surgery.

DETAILED DESCRIPTION:
LSG is defined as first-line bariatric surgery for patients at high surgical risk with better surgical outcomes. Effective postoperative pain management is essential for early mobilization, and reduction of the risk of morbidity and mortality. Opioids, due to their potent analgesic effects are used as a component of multimodal analgesia in the postoperative period. Despite their advantages, opioids may be related to pulmonary complications such as atelectasis and impaired alveolar gas exchange, apnea; postoperative delayed recovery due to ileus, nausea, and vomiting; and prolonged hospital stay. The use of interfascial plane blocks for pain management has increased recently, as ultrasonography (USG) has become a part of daily routine. Interfascial plane blocks provide effective postoperative analgesia.

Additionally, reducing postoperative opioid consumption helps to provide hemodynamic stability and promote early mobilization. Studies are showing M-TAPA block to be effective for postoperative analgesia for abdominal surgeries, and some studies continued comparing its effect in laparoscopic sleeve gastrectomy with other plane blocks. There are also case reports showing the effectiveness of the M-TAPA block in LSG patients. M-TAPA block's effect on LSG patients has not been studied yet. The investigators hypothesize that the M-TAPA block performed in patients undergoing laparoscopic sleeve gastrectomy would reduce opioid consumption in the first 24-hour period after surgery.

ELIGIBILITY:
Inclusion Criteria: American Society of Anesthesiologists (ASA) classification II- III Patients Scheduled for LSG under general anesthesia

-

Exclusion Criteria: Patients

* with a history of bleeding diathesis,
* receiving anticoagulant treatment,
* with allergies or sensitivity to drugs used,
* with an infection on the puncture site
* with a history of alcohol or drug addiction,
* with congestive heart failure
* with liver or kidney disease
* who do not accept the procedure or participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Opioid consumption | Changes from baseline opioid consumption at postoperative 0, 2, 4, 8, 16, and 24 hours
  The primary aim is to compare postoperative opioid consumption from the PCA device.

SECONDARY OUTCOMES:
Pain scores | Changes from baseline pain scores at postoperative 0, 2, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the Numerical Rating Scale (NRS) (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded.
Need for rescue analgesia (tramadol) | Postoperative 24-hour period
  The secondary aim is to compare rescue analgesia amount used in the postoperative 24 h period.
Adverse events | Postoperative 24-hour period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching, ect) related to opioid use

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Mega Hospital Complex, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share individual patient data (IPD).

REFERENCES:
- [Background] Schug SA, Raymann A. Postoperative pain management of the obese patient. Best Pract Res Clin Anaesthesiol. 2011 Mar;25(1):73-81. doi: 10.1016/j.bpa.2010.12.001. PMID 21516915
- [Result] Jackson TD, Hutter MM. Morbidity and effectiveness of laparoscopic sleeve gastrectomy, adjustable gastric band, and gastric bypass for morbid obesity. Adv Surg. 2012;46:255-68. doi: 10.1016/j.yasu.2012.05.002. PMID 22873044
- [Result] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Result] Tulgar S, Selvi O, Thomas DT, Deveci U, Ozer Z. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides effective analgesia in abdominal surgery and is a choice for opioid sparing anesthesia. J Clin Anesth. 2019 Aug;55:109. doi: 10.1016/j.jclinane.2019.01.003. Epub 2019 Jan 9. No abstract available. PMID 30639940
- [Result] Ciftci B, Gungor H, Alver S, Akin AN, Ozdenkaya Y, Tulgar S. Clinical Experience for Modified Thoracoabdominal Nerve Block Through Perichondrial Approach (M-TAPA) in Five Patients. Dermatomal Evaluation and Application of Different Volumes: A Case Series and Review of Literature. Turk J Anaesthesiol Reanim. 2023 Aug 18;51(4):354-357. doi: 10.4274/TJAR.2022.221042. PMID 37587679
- [Result] Aikawa K, Tanaka N, Morimoto Y. Modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) provides a sufficient postoperative analgesia for laparoscopic sleeve gastrectomy. J Clin Anesth. 2020 Feb;59:44-45. doi: 10.1016/j.jclinane.2019.06.020. Epub 2019 Jun 15. No abstract available. PMID 31212124